CLINICAL TRIAL: NCT05721378
Title: (Cost-)effectiveness of Permissive Weight Bearing in Surgically Treated Trauma Patients with Displaced Intra-Articular Calcaneal Fractures: a Multicenter, Randomized Controlled Trial
Brief Title: Permissive Weight Bearing in Displaced Intra-articular Calcaneal Fractures
Acronym: PIONEER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PIONEER
Record Dates: First submitted 2023-01-13; First posted 2023-02-10 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Calcaneus Fracture; Displaced Intra-Articular Fracture of Calcaneus (Diagnosis); Trauma Injury
Keywords: Permissive Weight Bearing; Rehabilitation
MeSH Terms: conditions — Disease; Accidental Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Permissive Weight Bearing group (Experimental): Rehabilitation following the Permissive Weight Bearing (PWB) protocol
  Interventions: Procedure: Permissive Weight Bearing group
- Restrictive Weight Bearing group (Active Comparator): Rehabilitation following the Restrictive Weight Bearing (RWB) protocol
  Interventions: Procedure: Restricted Weight Bearing group

INTERVENTIONS:
Procedure: Permissive Weight Bearing group — The Permissive Weight Bearing (PWB) protocol allows earlier post-operative permissive weight bearing, where progression of weight bearing is guided by the subjective experience (for example: pain, weight bearing tolerance) of the patient and the clinical expertise of the treating physician and therapist. Patients allocated to the PWB protocol start weight bearing after wound healing is achieved (approximately two weeks after the operation). Consequently, patients are stimulated to bear as much weight as tolerated by pain and comfort. Treatment will take place according to the PROMETHEUS protocol (treatment- and evaluation protocol). The protocol contains a number of weight bearing milestones (e.g. walking with two crutches, walking with two canes, walking with one cane and walking without any walking aids). The treating physiotherapist or physician records the dates that these milestones are reached in the study database.
  Other Names: Early Weight Bearing
  Arms: Permissive Weight Bearing group
Procedure: Restricted Weight Bearing group — The Restrictive Weight Bearing (RWB) protocol consists of 8 to 12 weeks of postoperative restricted weight (0-10%) bearing, following the current AO Guidelines (7). After 8 weeks of restricted weight bearing, the weight bearing will be increased with 25% per week for 4 weeks. Every time the patient and the treating physical therapist or physician have contact, the weight bearing advice given to the patient at that point in time is recorded (unloaded; partial weight bearing + clarification; full weight bearing). Also, any additional advice given to the patient is recorded.
  Other Names: Non Weight Bearing
  Arms: Restrictive Weight Bearing group

SUMMARY:
The goal of the proposed study is to define the optimal rehabilitation for trauma patients with Displaced Intra-articular Calcaneal Fractures, either Permissive Weight Bearing (PWB) or Restricted Weight Bearing (RWB) regarding functional outcomes, health related quality of life, radiographical differences, cost-effectiveness and complications.

DETAILED DESCRIPTION:
Rationale: Of all fractures, 1-2% involve the calcaneus. Often surgical treatment is needed. Even after successful treatment it requires long rehabilitation with major impact on daily life and socio-economic aspects. Anatomic surgical restoration does not prevent gait disturbances or persistent foot pain. An adequate rehabilitation program is mandatory to maximize foot stability.

Objective: Evidence showing which rehabilitation protocol is best for both fracture healing and quality of life for patients with Displaced Intra-Articular Calcaneal Fractures (DIACFs) is mostly lacking. This study has the aim to answer the question whether surgically treated patients with DIACFs following the Permissive Weight Bearing protocol (PWB) have better functional outcomes compared to patients with Restricted Weight Bearing protocol after 12 weeks (RWB) measured with the American Orthopaedic Foot & Ankle Society (AOFAS) Score. The study hypothesizes that patients with DIACFs following the PWB protocol will have a better quality of life (HR-QOL) compared to patients who followed the RWB protocol.

The hypothesis is that there will be lower costs without any radiographic differences for surgically treated (irrespective of technique used) patients with DIACFs following a PWB protocol comparing to the current AO (Arbeitsgemeinschaft für Osteosynthesefragen) standard care: the RWB protocol.

Study design: Multi-center randomized controlled trial

Study population: Presence of surgically (extended lateral, sinus tarsi or percutaneous approach) fixed DIACFs classified as Sanders type II to IV, age 18-67 years (labor force). Patients must be able to understand and follow weight bearing instructions. Patients will only be included after written informed consent is obtained.

Groups (intervention and control): Patients with DIACFs will be randomly allocated to one of the rehabilitation protocols, either PWB or RWB.

Main study parameters/endpoints: Primary objective: functional outcome. Secondary outcomes: quality of life, differences in radiographic parameters, complications, cost effectiveness and differences in surgical techniques.

Nature and extent of the burden: The PWB protocol aims to restore weight bearing faster than RWB protocol in DIACFs. Early postoperative weight bearing poses the risk of increased complications, such as secondary displacement of the fracture or failure of fracture fixation. Previous analysis of this protocol in other lower extremity fractures has shown a safe complication rate, although data from prospective randomized trials in calcaneus fractures are lacking. Follow-up is standardized according to current trauma guidelines, namely at time points 2, 6, 12 weeks and 6 months. The radiation exposure will not be different from standard of care. Therefore, the burden for participants is considered minimal, with no significant health risks.

ELIGIBILITY:
Inclusion Criteria:

* Surgically treated trauma patients with isolated unilateral DIACFs, less than 6 weeks after trauma, Sanders type II-IV (14)
* Age between 18 and 67 years old (labor force)
* Being able to understand the questionnaires and measurement instructions
* Indication for open/closed reduction and internal fixation
* Written Informed Consent

Exclusion Criteria:

* Acute or existing amputation (upper limb, lower limb, feet)
* Open calcaneal fractures (excluding medial wound without compromising surgical approach)
* Bilateral fractures of the lower extremities
* Unable to comply to the PWB protocol due to pre-existing conditions of the arms and legs (e.g. unable to use crotches due to hemiparalysis)
* Severe non-fracture related comorbidity of the lower extremity
* Pre-existent immobility (loss of muscle function of one or both legs)
* Dependent in activities of daily living (e.g. due to dementia, Alzheimer, New York Heart Association class IV angina, heart failure or oxygen-dependent chronic obstructive pulmonary disease)
* Rheumatoid arthritis of the lower extremities
* Severe psychiatric comorbidities that lead to inability to comply with the treatment protocol
* Pathologic fractures (metastasis, secondary osteoporosis)
* Peripheral neuropathy and/or diabetes
* Alcohol- or drug abuse preventing adequate follow-up
* Primary indication for arthrodesis subtalar joint
* Two or more fractures of the upper and/or lower extremities

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in functional outcome as defined by the AOFAS questionnaire | 0, 2, 6, 12 weeks and 6 months post-surgery.
  The American Orthopaedic Foot & Ankle Society (AOFAS) score is a clinician-based score. It incorporates both subjective and objective information. Patients report their pain, and physicians assess alignment. It is designed for physicians to help standardize the assessment of patients and makes the results of this study comparable with previous data. Scores range from 0 to 100, with healthy foot and ankles receiving 100 points.

SECONDARY OUTCOMES:
Self-reported function with the Maryland Foot Score | 0, 2, 6, 12 weeks and 6 months post-surgery
  The MFS is an assessment for foot disorders, mainly consisting of the following items: pain, gait, functional activities, and cosmesis. The scale scores have a minimum of 0 points and a maximum of 100 points. A total score of <50 is considered as poor, 50-74 as fair, 75-89 as good, and 90-100 as excellent.
Activities of Daily Living (ADL) with LEFS | 0, 2, 6, 12 weeks and 6 months post-surgery
  The lower extremity functional scale (LEFS) is a questionnaire containing 20 questions about a person's ability to perform everyday tasks. The LEFS can be used by clinicians as a measure of patients' initial function, ongoing progress, and outcome, as well as to set functional goals. The LEFS can be used to evaluate the functional impairment of a patient with a disorder of one or both lower extremities. It can be used to monitor the patient over time and to evaluate the effectiveness of an intervention. The questionnaire consists of 80 points. The lower the score the greater the disability.
Health Related Quality of Life with EQ-5D-5L | 0, 2, 6, 12 weeks and 6 months post-surgery
  The EuroQol 5-Dimension, 5-Level Health Scale (EQ-5D-5L) is a self-administered questionnaire, which will be completed at baseline together with the cost questionnaire at the same moments (0, 2, 6, 12 weeks and 6 months). Both generic quality of life, as well as utilities, will be derived by means of the EQ-5D-5L, which will be administered both by the patients. The Dutch version of the EQ-5D-5L is chosen because it is a widely used quality of life instrument (nationally and internationally) and it is recommended by the Dutch guidelines.The EQ-5D-5L contains 5 dimensions of health-related quality of life, namely mobility, self-care, daily activities, pain/discomfort and depression/anxiety. Each dimension can be rated at five levels: no problems to major problems. The 5 dimensions can be summed into a health state.
Böhlers angle and posterior facet joint | Early postoperative (before first mobilization) and 6 months post-surgery
  Radiographic evaluation by a radiologist blinded for treatment allocation will be done at the same time intervals as the scheduled visits to the physician.
  To see if there is a difference in the alignment of Böhlers angle and posterior facet joint alignment (radiographically measured), a CT-scan will be performed early post-operatively (before first weight bearing) and after 6 months. Differences in the Böhlers angle and posterior joint alignment (Δ = CT6months - CTpost-op.) will be calculated. The normal degree for the Böhler angle varieties between 25° and 40°. An intra-articular step off or gap from less than 2mm of the posterior facet was considered as well-reduced.
Medical consumption with iMCQ | 0 weeks and 6 months post-surgery
  The iMTA Medical Consumption Questionnaire (iMCQ) measures health care utilization and is based on 29 questions. It is an instrument for measuring medical consumption and is related to frequently occurring contacts with health care providers. The iMCQ is a generic questionnaire. It is therefore not disease specific. The questions ask about health care related appointments patients had in the past period. In case the respondent had no appointments, the score '0' is noted.
Society costs with iPCQ | 0 weeks and 6 months post-surgery
  The iMTA Productivity Cost Questionnaire (iPCQ) measures productivity losses. The questionnaire is based on 12 questions. Questions 1 to 3 give information about the amount of paid work (in hours) and the number of days per week on which the respondent works. The latter provides insight into the average number of hours of work per working day of the respondent. This information is needed to calculate productivity loss costs.
  The questions about productivity losses form the following modules:
  * Absenteeism: absenteeism from paid work (questions 4 to 6)
  * Presenteeism: productivity losses during days worked (questions 7 to 9)
  * Productivity loss from unpaid work (questions 10 to 12). After completing the questionnaire the total amount of absenteeism can be calculated by multiplying the number of days absent and the number of hours per working day of the respondent.
  To calculate the costs of productivity losses, volumes are multiplied by unit cost prices.
Occurrence of complications | 6 and 12 weeks and 6 months post-surgery
  Most important complications, such as: wound infection, dislocation, non-union, - failure of osteosynthesis, postoperative arthritis

CONTACTS AND LOCATIONS:
Locations (11):
- Netherlands (11):
  - Amsterdam University Medical Center, Amsterdam
  - Rijnstate Hospital, Arnhem
  - Amphia Hospital, Breda
  - Catharina Hospital, Eindhoven
  - Groene Hart Hospital, Gouda
  - Maastricht University Medical Center +, Maastricht
  - Radboud University Medical Center, Nijmegen
  - Maasstad Hospital, Rotterdam
  - Zuyderland Medical Center, Sittard
  - Haaglanden Medical Center, The Hague
  - Elisabeth-Twee Steden Hospital, Tilburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Verstappen C, Driessen MLS, Kalmet PHS, Brandts L, Kimman M, Edwards M, Hermans E, Poeze M. Permissive weight bearing versus restrictive weight bearing in surgically treated trauma patients with displaced intra-articular calcaneal fractures (the PIONEER study): study protocol for a multicenter randomized controlled trial. Trials. 2024 Nov 18;25(1):778. doi: 10.1186/s13063-024-08617-5. PMID 39558368